CLINICAL TRIAL: NCT05863299
Title: Sleep Quality of Critically Ill Children Change Trajectory and Prediction Factors: A Prospective Longitudinal Mixed Study
Brief Title: A Prospective Longitudinal Mixed Study on the Change Track of Sleep Quality in Critically Ill Children
Status: Completed | Type: Observational
Sponsor: Children's Hospital of Fudan University (Other)
Responsible Party: Sponsor
Other Study IDs: CHFudanU
Record Dates: First submitted 2023-05-08; First posted 2023-05-18 (Actual); Last update posted 2024-02-07 (Actual); Status verified 2024-02

CONDITIONS: Critical Illness; Child; Sleep Disorder
MeSH Terms: conditions — Critical Illness; Sleep Wake Disorders

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
This research adopts the uniform parallel hybrid research design; The quantitative data and qualitative data were collected at the same time, and then the quantitative and qualitative data were analyzed respectively. Finally, the two data sets were combined. Comprehensive interpretation of the study issues through complementarity and mutual validation of quantitative and qualitative data.

DETAILED DESCRIPTION:
With the progress and development of medical technology, the mortality rate of critically ill children continues to decline. To improve the long-term prognosis of children has become a new goal of modern medicine. Sleep disorders in critically ill children are caused by disease factors, the complex environment of ICU, and various treatment factors, which have seriously affected the patient's rehabilitation and long-term quality of life. Attention should be paid to the sleep disorders in critically ill children. At present, the research on sleep disorders in critically ill patients in China is mostly focused on adults, and the critically ill children are rarely involved, and there is no research related to sleep disorders and recovery tracks of critically ill children. This prospective longitudinal mixed study aims to describe the change trajectory of sleep disorder and recovery in critically ill children and provide suggestions for subsequent clinical workers to formulate reasonable intervention measures.

ELIGIBILITY:
Inclusion Criteria:

① Age 3-12 years;

* Children who are conscious during ICU,
* children with Glasgow score of 15

Exclusion Criteria:

* (1) did not meet the discharge standards, and asked to be discharged;

  * Children with sleep disorder before admission to PICU, that is, those with baseline CSHQ score > 41;

    * The child had a history of mental illness and cognitive impairment.

      * Children with brain injury, coma, disturbance of consciousness, epilepsy and status epilepticus, obstructive sleep apnea hypopnea syndrome; ⑤ Children with hearing and hearing impairment ⑥ICU stay > 30 days.

Ages: 2 Years to 16 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: 3-12 years chlidren who are conscious in ICU
Sampling Method: Probability Sample
Enrollment: 247 (Actual)
Dates: Start 2022-11-17 (Actual); Primary Completion 2023-12-17 (Actual); Study Completion 2023-12-31 (Actual)

PRIMARY OUTCOMES:
Mean Total Night Sleep Minutes | 2023.12.31
  Mean Total Night Sleep Minutes
Deep sleep time | 2023.12.31
  Deep sleep time
Children sleep habit questionnaire score | 2023.12.31
  Children sleep habit questionnaire score

CONTACTS AND LOCATIONS:
Overall Officials: Ying Gu, Study Chair — Pediatric Hospital Affiliated to Fudan University
Locations (1):
- Children's Hospital of Fudan University, Shanghai, China

IPD SHARING:
Plan to Share IPD: Undecided